CLINICAL TRIAL: NCT01465789
Title: Noninvasive Biomarkers for Monitoring Cardiometabolic Risk in Children
Status: Terminated | Type: Observational
Why Stopped: Loss of participants to follow-up
Sponsor: West Virginia School of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Kristie Bridges, Associate Professor, West Virginia School of Osteopathic Medicine
Other Study IDs: BCS 102.2
Record Dates: First submitted 2011-07-05; First posted 2011-11-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify salivary biomarkers for monitoring cardiometabolic risk in children. The study hypothesis is that a combination of salivary biomarkers will predict the presence of risk factors including impaired fasting glucose, hypertension and dyslipidemia and will reflect changes in these risk factors over time.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the CARDIAC Boot Camp Program
* Between the ages of 4 and 17
* Parental permission
* Ability to provide assent

Exclusion Criteria:

* Inability to comply with saliva collection procedures
* Renal insufficiency or juvenile gout

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children participating in the CARDIAC Boot Camp program at the Robert C. Byrd Clinic in Lewisburg WV
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Correlation (R values) of salivary biomarkers with blood pressure percentile and serum glucose, HDL, total cholesterol, triglyceride and insulin levels in children | Baseline
Predictive utility (C-statistic) of salivary biomarkers for development of metabolic syndrome during childhood and adolescence | final assessment at age 18 (up to 14 years depending on age of enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie G Bridges, PhD, Principal Investigator — West Virginia School of Osteopathic Medicine; Jill Cochran, PhD, MSN, RN-C FNP, Principal Investigator — West Virginia School of Osteopathic Medicine
Locations (1):
- West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia, United States